CLINICAL TRIAL: NCT05012774
Title: Speech Perception Training: Advanced Scoring and Feedback Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SeeHear LLC (Industry)
Collaborators: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DC015418
Record Dates: First submitted 2021-08-02; First posted 2021-08-19 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Hearing Loss
Keywords: lipreading speechreading; perceptual learning; adults with acquired hearing loss; multisensory speech processing; remote training system; speech recognition in noise; perceptual feedback during training
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: In Aim 1, which is sentence lipreading training, the intervention compares the provision of three different types of feedback for lipreading. The three types are consonant-level, word-level, or sentence-level feedback. A no-training wait-list control is included.
  In Aim 2, novel word training, the intervention has one arm in which novel word learning via lipreading the words is supported by allowing the participants to read the consonants in the novel words before lipreading them.
  In Aim 3, the most effective feedback with sentence training will be compared with novel word training using training stimuli that are audiovisual speech in speech-shaped noise.
  The interventions are all delivered individually via the web. Finally, all pre- and post-training results will be compared across groups including the wait-list controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Aim 1, Sentence Training: Sentence Feedback (Experimental): In Aim 1, which is sentence lipreading training, the intervention compares the provision of three different types of feedback for lipreading.
  This arm gives printed whole sentence feedback following an attempt to lipread each sentence.
  Participants receive pre- and post-training tests.
  Interventions: Behavioral: Speech Recognition Training
- Aim 1, Sentence Training: Word Feedback (Experimental): In Aim 1, which is sentence lipreading training, the intervention compares the provision of three different types of feedback for lipreading.
  This arm gives printed whole word feedback following an attempt to lipread each sentence. Word feedback is for correct words and words that are perceptually similar but incorrect responses.
  Participants receive pre- and post-training tests.
  Interventions: Behavioral: Speech Recognition Training
- Aim 1, Sentence Training: Consonant Feedback (Experimental): In Aim 1, which is sentence lipreading training, the intervention compares the provision of three different types of feedback for lipreading.
  This arm gives printed consonant word feedback following an attempt to lipread each sentence. Word feedback is for correct words, but only the consonants are given as feedback for words that are perceptually similar but incorrect responses.
  Participants receive pre- and post-training tests.
  Interventions: Behavioral: Speech Recognition Training
- Aim 1, Sentence Training: No Training Control (No Intervention): Participants receive only the pre- and post-training tests.
- Aim 2, Nonsense Word Training (Experimental): Participants train to lipread nonsense words that name nonsense pictures. Participants receive pre- and post-training tests.
  Interventions: Behavioral: Speech Recognition Training
- Aim 3, Audiovisual Nonsense Word Training (Experimental): Participants train to recognize audiovisual spoken nonsense words that name nonsense pictures and are presented in speech-shaped noise. The paradigm is the same as in Aim 2.
  Participants receive pre- and post-training tests.
  Interventions: Behavioral: Speech Recognition Training
- Aim 3, Audiovisual Sentence Training (Experimental): Participants receive the same training paradigm from Aim 1 with the most effective feedback type from Aim 1. But the sentences are audiovisual and in speech-shaped noise.
  Participants receive pre- and post-training tests.
  Interventions: Behavioral: Speech Recognition Training

INTERVENTIONS:
Behavioral: Speech Recognition Training — Training for each training arm takes place over 10 sessions carried out at home. on the participant's own computer without experimenter direct supervision. Pre- and post-training tests are carried out under experimenter supervision.
  Arms: Aim 1, Sentence Training: Consonant Feedback; Aim 1, Sentence Training: Sentence Feedback; Aim 1, Sentence Training: Word Feedback; Aim 2, Nonsense Word Training; Aim 3, Audiovisual Nonsense Word Training; Aim 3, Audiovisual Sentence Training

SUMMARY:
The purpose of the study is to assess training of visual speech (lipreading) and audiovisual (lipreading plus auditory) speech as a rehabilitation strategy for hearing loss in adults.

DETAILED DESCRIPTION:
It is hypothesized that training that improves lipreading in older adults can carry over to untrained lipreading materials and to audiovisual speech recognition in noise. Participants receive pre- and post-training tests of speech recognition with visual-only, auditory-only, and audiovisual spoken sentences and isolated words. During pre- and post-training tests, they carry out forced choice identification of lipread consonants. Participants who are assigned to a training arm train on lipreading isolated sentences (Aim 1) or on learning via lipreading sets of isolated nonsense words (Aim 2). Depending on the outcomes of Aims 1 and 2, in Aim 3, new participants receive audiovisual training with conditions from Aims 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Must have Mild to severe hearing loss
* Native speaker of American English
* Access to computer and the ability to use it for the testing, training, and teleconferencing
* computer display >= 10 inches diagonal

Exclusion Criteria:

* Internet too slow for streaming
* History of brain trauma or learning disability
* Poor (corrected) vision

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in words-correct scores across pre- and post-training sentence lipreading tests. | up to 8 weeks
  Change in words-correct scores across pre- and post-training visual-only sentence tests with open-set responses.
Change in phonemes-correct scores across pre- and post-training sentence lipreading tests. | up to 8 weeks
  Change in phonemes-correct scores across pre- and post-training visual-only sentence tests with open-set responses.
Change in consonant-identification scores across pre- and post-training word lipreading tests. | up to 8 weeks
  Change in consonants-correct scores across pre- and post-training for visual-only tests using isolated nonsense words and closed-set responses.
Change in word-correct scores across pre- and post-training word lipreading tests. | up to 8 weeks
  Change in words-correct scores across pre- and post-training visual-only isolated real word tests with open-set response.
Change in phonemes-correct scores across pre- and post-training word lipreading tests. | up to 8 weeks
  Change in phonemes-correct scores across pre- and post-training visual-only isolated real word tests with open-set response.

SECONDARY OUTCOMES:
Change in words-correct scores across pre- and post-training audiovisual sentence tests. | up to 8 weeks
  Change in words-correct scores across pre- and post-training audiovisual-in-noise sentence identification tests with open-set response.
Change in phonemes-correct scores across pre- and post-training audiovisual sentence tests. | up to 8 weeks
  Change in phonemes-correct scores across pre- and post-training audiovisual-in-noise sentence identification tests with open-set response.
Change in word-correct scores across pre- and post-training for audiovisual-in-noise word tests. | up to 8 weeks
  Change in word-correct scores across pre- and post-training audiovisual-in-noise isolated real word tests with open-set response.
Change in phoneme-recognition scores across pre- and post-training audiovisual-in-noise word tests. | up to 8 weeks
  Change in phoneme-recognition scores across pre- and post-training audiovisual-in-noise isolated real word tests with open-set response.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne E Bernstein, Ph.D., Study Director — George Washington University
Locations (1):
- George Washington University, Washington, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with other researchers following appropriate agreements. Personally-identifiable data will never be shared with individuals outside the research team, except as required by Law, NIH, or Geourge Washington University.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after they have been described in publications by the authors.
Access Criteria: The data will be transferred via the Open Science Framework.
URL: http://osf.org

DOCUMENTS (1):
  • Informed Consent Form (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT05012774/ICF_000.pdf